CLINICAL TRIAL: NCT02191982
Title: A Randomized, Wait-list Controlled Clinical Trial: the Effect of a Physical Activity Program on Fatigue After Potentially Curative Chemotherapy Among Cancer Survivors Age 65 or Older -- PACT (Physical Activity After Chemotherapy)
Brief Title: The Effect of Walking on Fatigue After Chemotherapy in Patients 65 and Older
Acronym: S-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1402
Record Dates: First submitted 2014-06-20; First posted 2014-07-16 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Cancer; Geriatric; Fatigue
Keywords: Cancer; Chemotherapy; Fatigue; Elderly; Geriatric; Any Cancer; Cancer Treatment; Weakness; Tiredness
MeSH Terms: conditions — Neoplasms; Fatigue; Asthenia | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This arm will begin the Walk With Ease program after the completion of chemotherapy.
  Interventions: Behavioral: Walk With Ease
- Wait List Control (Active Comparator): The arm will begin the Walk With Ease program three months after completion of chemotherapy.
  Interventions: Behavioral: Walk With Ease

INTERVENTIONS:
Behavioral: Walk With Ease — Walk With Ease is the Arthritis Foundation's evidence-based walking intervention to help with fatigue and pain. The intervention is a self-directed program that helps guide participants in a safe and comfortable paced walking program with an ultimate goal of walking for 30 minutes a day, five days a week.
  Other Names: WWE

SUMMARY:
This study will look at the impact of a self-directed walking program on post-chemotherapy survivors experiencing fatigue. It is hypothesized that the walking program will help lessen fatigue.

DETAILED DESCRIPTION:
The investiagors propose to evaluate the impact of a home-based self-directed walking program on post-chemotherapy fatigue among 150 cancer survivors age 65 and older -- Senior Physical Activity after Chemotherapy (S-PACT). Participants must have potentially curable cancer, moderate to severe fatigue (score of 4 or higher on the Brief Fatigue Inventory), currently exercise less than 120 minutes per week and have completed chemotherapy treatment (radiation treatment must also be completed if it is part of the patient's treatment plan) within the last 6 weeks. The design is a randomized controlled trial, with participants randomized to a 3-month physical activity program (intervention group) or to wait-list control (this group begins the walking program at 3 months post-randomization). The primary objective is to compare the change in fatigue scores from baseline to 3 months between the intervention and wait-list control groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 65 years and older
* Histologically or cytologically confirmed cancer (hematologic or solid) at stage considered amenable to cure as assessed by the treating MD
* Within 6 weeks of end of chemotherapy (all participants must have had chemotherapy treatment)

  * Any radiation received must also be completed prior to randomization (if radiation treatment follows adjuvant chemotherapy, then the patient must be recruited within 6 weeks of end of radiation)
  * Maintenance hormonal therapy in women with breast cancer is allowed; see exclusion criteria regarding hormonal therapy in males with prostate cancer
* Moderate to severe fatigue (>4 on BFI)
* Less than 120 minutes/week of physical activity
* English speaking
* Signed IRB approved written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements.

Exclusion Criteria:

* Receiving hormonal therapy for prostate cancer
* Unable to walk or engage in moderate-intensity physical activity
* Have BFI≤3.
* Report more than 120 minutes/week of physical activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To measure change in fatigue scores between intervention and wait list control arms from baseline to three months. | Three months
  Change in fatigue will be measured using the FACIT-F.

SECONDARY OUTCOMES:
To measure change in fatigue scores between intervention and WLC arms from baseline to 3 months | Three months
  This outcome will be measured by the Brief Fatigue Inventory
To report recruitment and retention in the study at 3 months | Three months
To report recruitment and retention in the study at 6 months | Six months
To measure implementation of and adherence to WWE | Six months
To count the number of adverse events | Six months
  To characterize the safety of the walking program through a review of the number and type of adverse events, including falls, reported by study participants to the Study Team.
To measure change in engagement of walking over time from baseline to three months. | Three Months
  To evaluate the following measures at baseline and 3 months, and compare changes in these measures over time between intervention and WLC arms.
  Engagement in walking (total minutes per week) as measured by engagement in physical activity questions
To measure change in physical function over time from baseline to three months. | Three Months
  To evaluate the following measures at baseline and 3 months, and compare changes in these measures over time between intervention and WLC arms.
  Physical function as measured by SPPB
To measure change in quality of life over time from baseline to three months. | Three Months
  To evaluate the following measures at baseline and 3 months, and compare changes in these measures over time between intervention and WLC arms.
  Quality of life as measured by FACT-G (global and subscales) and symptom scales, including PROMIS pain intensity, sleep disturbance and depression.
To measure change in self-efficacy over time from baseline to three months. | Three Months
  To evaluate the following measures at baseline and 3 months, and compare changes in these measures over time between intervention and WLC arms.
  Engagement in walking (total minutes per week) as measured by engagement in physical activity questions

CONTACTS AND LOCATIONS:
Overall Officials: Hyman B Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Geriatric Oncology Program — https://unclineberger.org/patientcare/programs/geriatric